CLINICAL TRIAL: NCT02538965
Title: A Phase 2, Multicenter, Single-arm, Open-label Study to Evaluate the Activity, Safety and Pharmacokinetics of Lenalidomide (Revlimid®) in Pediatric Subjects From 1 to = 18 Years of Age With Relapsed or Refractory Acute Myeloid Leukemia.
Brief Title: A Study of Lenalidomide in Pediatric Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-AML-002
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Leukemia, Myeloid
Keywords: Lenalidomide; Revlimid; Pediatric; Relapsed or Refractory; Acute Myeloid Leukemia; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid; Recurrence; Leukemia, Myeloid, Acute; Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide API will administered at a starting dose of 2 mg/kg/day. Lenalidomide will be provided as either a capsule (2.5 mg, 5 mg, 10 mg, 15 mg, 20 mg or 25 mg) or as an oral suspension (10mg/mL).
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide will be administered orally once daily for the first 21 days of every 28-day cycle. The starting dose will be 2 mg/kg/day with a maximum dose of 70 mg/day. Number of cycles: 12, or until evidence of progressive disease. Participants will also be discontinued if unresolved toxicities as described in the protocol occur, or if dose reductions are required and subject does not tolerate minimum dose level of 1mg/kg/day.

SUMMARY:
To determine the activity of lenalidomide in the treatment of pediatric subjects with relapsed/refractory acute myeloid leukemia (AML) (with second or greater relapse or refractory to at least 2 prior induction attempts) measured by morphological complete response defined as either a CR or CRi within the first 4 cycles of treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, Phase 2, Simon's Optimal two-stage design study, with an Optional Extension Phase (OEP), that will assess the activity, safety and pharmacokinetics (PK) of lenalidomide in pediatric subjects from 1 to ≤ 18 years of age with second or greater Relapsed or Refractory Acute Myeloid Leukemia (rrAML). A total of 43 evaluable participants (18 participants in Stage 1 and an additional 25 participants in Stage 2) are required for assessment of the primary endpoint. To allow for participants found to be unevaluable for the primary endpoint due to an incorrect diagnosis, not having a disease assessment post screening, or who discontinued prior to receiving lenalidomide, up to 4 additional participants may be enrolled for a maximum of 47 evaluable subjects across approximately 70 sites. Approximately 50% of enrolled participants will be younger than 12 years of age to provide adequate PK data for this age subset.

If during Stage 1, at least 3 of 18 participants achieve a morphologic complete response (either CR or CRi) within the first 4 cycles of study treatment, then the study will proceed to Stage 2; otherwise, the study will be terminated. Similarly, if at the final analysis, at least 8 of 43 evaluable subjects across Stages 1 and 2 achieve a response (CR/CRi) within the first 4 cycles of study treatment, it will be concluded that lenalidomide has sufficient activity in pediatric Acute Myeloid Leukemia (AML) to warrant subsequent study. The optional extension phase (OEP) will allow participants who demonstrate clinical benefit, as assessed by the Investigator at the completion of 12 cycles of lenalidomide therapy, to continue receiving oral lenalidomide until they meet the criteria for study discontinuation. In the OEP, only safety, dosing, concomitant medications/procedures, and second primary malignancies (SPMs) will be monitored.

ELIGIBILITY:
Inclusion Criteria:

- Participants must satisfy the following criteria to be enrolled in the study:

1. Male or female is 1 to ≤ 18 years of age at the time of signing the Informed Consent Form / Informed Assent Form (ICF/IAF).
2. Participants (when applicable, parental/legal representative) must understand and voluntarily provide permission to the ICF/IAF prior to conducting any study-related assessments/procedures.
3. Participants have relapsed or refractory acute myeloid leukemia after at least 2 prior induction attempts:

   * Bone marrow aspirate or biopsy must have ≥ 5% blasts by morphology and/or flow cytometry.
   * Each block of chemotherapy is a separate reinduction attempt.
   * Donor lymphocyte infusion (DLI) is considered a reinduction attempt.
4. Participants are willing and able to adhere to the study visit schedule and other protocol requirements.
5. Participants have a Karnofsky score of ≥ 50% (participants ≥ 16 years of age) or a Lansky score ≥ 50% (participants < 16 years of age).
6. Participants have a resting left ventricular ejection fraction (LVEF) of ≥ 40% obtained by echocardiography.
7. Participants have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to first dose. All prior treatment-related toxicities must have resolved to ≤ Grade 2 prior to enrollment.
8. Regarding radiation therapy, time elapsed prior to first dose of lenalidomide:

   * 2 weeks for local palliative radiation therapy (XRT).
   * 8 weeks if prior craniospinal chemoradiation therapy (CRT) or if ≥ 50% radiation of pelvis.
   * 6 weeks if other bone marrow radiation has been administered.
9. Graft-versus-host disease criteria:

   * Participants must be at least 2 months (from first dose of lenalidomide) from stem cell infusion.
   * Participants must have no evidence of active acute or chronic GVHD (Grade 0) for 4 weeks prior to the first dose of lenalidomide.
   * If the participants have a history of maximum Grade 1 or 2 GVHD that was treated with systemic steroid (≥ 0.5 mg/kg/day prednisone equivalents) or other non-steroid systemic IST, the participant must be off all IST for at least 2 weeks, and must have ceased treatment doses of steroids for GVHD (≥ 0.5 mg/kg/day prednisone equivalents) for at least 4 weeks.

     * If the participants have a history of Grade 3 or greater GVHD, the participants must be off all systemic IST for 4 weeks
     * Topical therapy is permitted and does not imply the participants have active acute or chronic GVHD.
   * Physiologic dosing of hydrocortisone is permitted.
10. At least 4 weeks (from first dose) elapsed from donor lymphocyte infusion (DLI) without conditioning.
11. Participants have adequate renal function, which is defined as:

    - Creatinine clearance calculated using the Schwartz formula, or radioisotope glomerular filtration rate (GFR) > 70 mL/min/1.73 m2.
12. Participants have adequate liver function, which is defined as:

    * Total bilirubin is ≤ 2 mg/dL unless the increase in bilirubin is attributable to Gilbert's Syndrome
    * Aspartate aminotransferase (AST) is ≤ 3.0 x upper normal limit (ULN) for age. For the purpose of this study, the ULN for AST is 50 U/L.
    * Alanine transaminase (ALT) is ≤ 3.0 x upper normal limit (ULN) for age. For the purpose of this study, the ULN for ALT is 45 U/L.
13. Female Children of Childbearing Potential (FCCBP), Female of Childbearing Potential (FCBP) and male participants that have reached puberty must agree to undergo physician-approved reproductive education and discuss the side effects of the study therapy on reproduction with parent(s) and/or guardian(s).
14. All participants and/or parents/guardians must have an understanding that lenalidomide could have a potential teratogenic risk. Female children of childbearing potential, is defined as females who have achieved menarche and/or breast development in Tanner Stage 2 or greater and have not undergone a hysterectomy or bilateral oophorectomy and FCBP defined as a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy and has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) must meet the following conditions below (Note: Amenorrhea following cancer therapy does not rule out childbearing potential):

    * Medically supervised serum pregnancy tests with a sensitivity of at least 25 mIU/mL must be conducted in FCCBP/FCBP, including those who commit to complete abstinence*. FCCBP/FCBP must have two pregnancy tests (with a minimum sensitivity of 25 mIU/mL) prior to starting treatment with lenalidomide. The first pregnancy test must be performed within 10 - 14 days prior to the start of lenalidomide treatment and the second pregnancy test must be performed within 24 hours prior to starting treatment with lenalidomide.

NOTE: The pregnancy test 10 to 14 days prior to initiation of lenalidomide may be omitted, at the discretion of the investigator, for any FCCBP/FCBP who has high acuity disease requiring immediate treatment with lenalidomide. The pregnancy test within 24 hours prior to the first dose of lenalidomide is required to be performed.

The participants may not received Investigational Product (IP) until the investigator has verified that the results of these pregnancy tests performed on Cycle 1 Day 1 are negative. FCCBP/FCBP with regular or no menstrual cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study Treatment Discontinuation Visit, and at Day 28 following IP discontinuation. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study Treatment Discontinuation Visit, and at Days 14 and 28 following IP discontinuation.

* Female participants must, as appropriate to age and at the discretion of the study Investigator, either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) and/or agree to the use of two reliable forms of approved and effective contraceptive methods simultaneously. The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) without interruption, 28 days prior to starting lenalidomide treatment, throughout the entire duration of study treatment including dose interruptions and 28 days after the end of study treatment.
* All male and female participants must follow all requirements defined in the Pregnancy Prevention Program.

  16. Male participants, as appropriate to age and the discretion of the study physician:
* Must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following lenalidomide discontinuation, even if he has undergone a successful vasectomy or practices complete abstinence.

Exclusion Criteria:

1. Participants have Down syndrome.
2. Participants have French-American-British classification (FAB) type M3 leukemia (acute promyelocytic leukemia) or identification of t(15;17).
3. Participants have isolated central nervous system (CNS) involvement or extramedullary relapse. (Participants with combined CNS/marrow relapse may be enrolled).
4. Participants had prior treatment with cytotoxic chemotherapy within 2 weeks of the first dose of lenalidomide with the exception of hydroxyurea (allowed prior to the first dose of lenalidomide and through Day 14 of Cycle 1) and intrathecal (IT) cytarabine will be administered within 2 weeks prior to administration of lenalidomide.
5. Participants have had prior treatment with biologic antineoplastic agents less than 7 days before the first dose of lenalidomide. For agents that have known adverse events (AEs) occurring beyond 7 days after administration (ie, monoclonal antibodies), this period must be extended beyond the time during which acute AEs are known to occur.
6. Participants have had prior treatment with lenalidomide.
7. Participant is pregnant or lactating.
8. Participants have an uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
9. Participants has known Human Immunodeficiency Virus (HIV) positivity (participants who are receiving antiretroviral therapy for HIV disease).
10. Participants have a prior history of malignancies other than AML unless the subject has been free of the disease for ≥ 5 years from first dose of lenalidomide.
11. The presence of any of the following will exclude a participant from enrollment:

    * Participants have any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
    * Participants have any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.
    * Participants have any condition that confounds the ability to interpret data from the study.
12. Participants have cardiac disorders (Common Terminology Criteria for Adverse Events [CTCAE] version 4.03 Grade 3 or 4).
13. Participants have a history of well-documented prior veno-occlusive disease (VOD).
14. Participants have any other organ dysfunction (CTCAE version 4.03 Grade 4) that will interfere with the administration of the therapy according to this protocol.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bouchra Benettaib, MD, Study Director — Celgene Corporation
Locations (62):
- United States (56):
  - Children's Hospital, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - Loma Linda University, San Bernardino, California
  - UCSF Children's Hospital, San Francisco, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I Dupont Hospital For Children, Wilmington, Delaware
  - Children's Hospital National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Advocate Chilldren's Hospital, Oak Lawn, Illinois
  - Riley Hospital For Children at IU Health, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Specialty Center of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hosp, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Inst, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Carolinas Healthcare System, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (6):
  - Alberta Childrens Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Center, Halifax, Nova Scotia
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec
  - Hospital For Sick Children, Torento

REFERENCES:
- [Derived] O'Brien MM, Alonzo TA, Cooper TM, Levine JE, Brown PA, Slone T, August KJ, Benettaib B, Biserna N, Poon J, Patturajan M, Chen N, Simcock M, Zimmerman L, Kolb EA. Results of a phase 2, multicenter, single-arm, open-label study of lenalidomide in pediatric patients with relapsed or refractory acute myeloid leukemia. Pediatr Blood Cancer. 2021 Jul;68(7):e28946. doi: 10.1002/pbc.28946. Epub 2021 Mar 10. PMID 33694257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 15 centers within the United States and Canada.
Pre-assignment Details: The study population consisted of pediatric participants with relapsed or refractory Acute Myeloid Leukemia (rrAML) from 1 to ≤ 18 years of age and were required to have a fresh bone marrow aspirate and biopsy submitted for confirmation of disease.
Groups:
- Lenalidomide: Participants received oral lenalidomide (capsules or suspension) at 2 mg/kg/day with a maximum dose of 70 mg/day for the first 21 days of each 28-day treatment cycle up to a maximum of 12 cycles of study treatment unless there was the development of a toxicity or adverse event (AE), death, withdrawal by parent/guardian of participant, lost to follow-up, pregnancy, non-compliance with investigational product (IP), physician decision, protocol violation or other reason. Upon completion or discontinuation of study treatment, participants entered the follow-up period for up to 5 years.
Period: Treatment Period
Arm/Group | Lenalidomide
Started | 17
Completed | 0
Not Completed | 17
Not completed — Other = Death due to disease progression | 1
Not completed — Adverse Event | 2
Not completed — Withdrawal by Parent/Guardian | 2
Not completed — Treatment Failure | 9
Not completed — Disease Progression | 1
Not completed — Physician Decision | 2
Period: Follow-Up Period
Arm/Group | Lenalidomide
Started | 17
Completed | 0
Not Completed | 17
Not completed — Other = Death due to disease progression | 13
Not completed — Withdrawal by Parent | 4

BASELINE CHARACTERISTICS:
Population: The intention to treat (ITT) population consisted of all enrolled participants regardless of whether they received lenalidomide.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (4.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 0
  White | 12
  Not Collected or Reported | 3
  Other | 1
Age Categories [Count of Participants; unit: Participants]
  ≤ 2 years | 0
  3-6 years | 4
  7-12 years | 6
  13-16 years | 4
  ≥ 17 years | 3
Peripheral Blood Smear Blasts [Median (Full Range); unit: Percent of Blasts] — Laboratory results obtained at baseline/screening include the peripheral white blood cells and blast counts, bone marrow blast percentage, cytogenetics and molecular alterations. Population: Includes participants with available data.
  Percent of Blasts
    number analyzed (Participants) | 15
    (all) | 8.7 [0 to 91]
White Blood Cell Count [Median (Full Range); unit: 10^9/L] — Laboratory results obtained at baseline/screening include the peripheral white blood cells and blast counts, bone marrow blast percentage, cytogenetics and molecular alterations.
  10^9/L | 3.700 [0.13 to 158.90]
Bone Marrow (BM) Myeloblasts Count [Median (Full Range); unit: Percent of Myeloblasts] — Laboratory results obtained at baseline/screening include the peripheral white blood cells and blast counts, bone marrow blast percentage, cytogenetics and molecular alterations. Population: Participants with available data.
  Percent of Myeloblasts
    number analyzed (Participants) | 16
    (all) | 57.5 [7 to 92]
Number of Participants With at Least One Cytogenetic Abnormality [Count of Participants; unit: Participants] — A standard cytogenetic metaphase preparation from the fresh bone marrow aspirate was prepared for the cytogenetic testing/chromosome analysis including karyotype. Results from cytogenetics, FISH studies, flow cytometry studies, and molecular studies performed locally at initial diagnosis and/or relapse was reported for t(16;16), t(8;21), MLL (11q23), t(15;17), monosomy 7, del(5q), or any other recurring abnormalities and presence or absence of mutations. More than one category can apply to a participant.
  Participants
    t(8;21) | 1
    +8 | 1
    complex (>/= 3 abnormalities) | 5
    -7 | 1
    7q- | 2
    11q 23 abnormalities | 3
    inv (3) | 1
    Other | 9
Number of Prior Systemic Anti-Cancer Regimens [Median (Full Range); unit: regimens] | 5 [2 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Morphologic Complete Response Within the First Four Cycles of Lenalidomide Treatment According to the Modified International Working Group (IWG) Criteria
Description: The morphological complete response rate was defined as the total number of participants with morphological CR observed within the first 4 cycles of lenalidomide (regardless of whether the CR/CRi was observed at the end of Cycle 1, 2, 3 or 4) over the total number of participants evaluable for this endpoint. According to Modified IWG criteria, morphologic CR was defined as:
  1. Absolute neutrophil count (ANC) ≥ 1000/μL and platelets ≥ 100,000 without transfusions and/or exogenous growth factor support (i.e., no transfusion or exogenous growth factor within 7 days of assessment;
  2. Bone marrow < 5% blasts evidence of trilineage hematopoiesis;
  3. No evidence of extramedullary disease.
  Morphologic CRi was defined as:
  1. ANC < 1000/μL and platelets < 100,000/μL or > 100,000/μL without platelet recovery (requiring transfusion within 7 days of assessment);
  2. BM with < 5% blasts and evidence of trilineage hematopoiesis;
  3. No evidence of extramedullary disease.
Time Frame: From day of the first dose of IP to end of cycle 4; Response was assessed at the completion of the 21-day treatment period of cycles 1, 2, 3, and 4 and at treatment discontinuation.
Population: The Intent to Treat (ITT) population consisted of all enrolled participants regardless of whether they received lenalidomide. Analysis was not completed due to scarcity of relevant data. See description.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Participants | 1 [0.1 to 28.7]

2. Secondary Outcome: Number of Participants Who Achieved a Bone Marrow Confirmed CR/CRi Lasting 3 Months (Durable Response Rate)
Description: Durable response rate was defined as the percentage of participants who achieved a BM confirmed CR/CRi according to the Modified IWG Response Assessment Lasting 3 Months (from the time to complete response observed until treatment failure or worse) or until transplantation if earlier among all participants eligible for durable response rate analysis, provided the CR/CRi was confirmed in a bone marrow sample). Due to scarcity of relevant data, it was not practical or meaningful to analyze the durable response rate. Only 1 participant had a response and the participant was censored soon after, as the consent was withdrawn; unable to calculate duration of response.
Time Frame: From date of confirmed complete response observed until treatment failure or worse; up to data cut-off date of 31 December 2017
Population: Due to scarcity of relevant data, it was not practical or meaningful to analyze the durable response rate. See description.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from date of the first observed response (CR, CRi or PR) until morphologic relapse, molecular/cytogenetic relapse, or death only for participants who achieved a response. Due to scarcity of relevant data, it was not practical or meaningful to analyze the duration of response. Only 1 participant had a response and the participant was censored soon after, as the consent was withdrawn; unable to calculate duration of response.
Time Frame: From date of first time of complete response observed until treatment failure or worse; up to data cut-off date of 31 December 2017
Population: ITT population participants that achieved at least a CR or CRi.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants Who Achieved a Best Response of Morphologic Complete Remission, Morphologic Complete Remission Incomplete or Partial Remission
Description: Overall response rate was defined as the number of participants with best response of CR, CRi or PR.
  A CR was defined as:
  1. ANC ≥ 1000/μL and platelets ≥ 100,000 without transfusions and/or exogenous growth factor support (no transfusion or exogenous growth factor within 7 days of assessment);
  2. BM < 5% blasts evidence of trilineage hematopoiesis;
  3. No evidence of extramedullary disease.
  A CRi was defined as:
  1. ANC < 1000/μL and platelets < 100,000/μL or > 100,000/μL without platelet recovery (requiring transfusion within 7 days of assessment);
  2. BM with < 5% blasts and evidence of trilineage hematopoiesis;
  3. No evidence of extramedullary disease.
  A PR was defined as:
  1. ANC of ≥ 1000/μL and platelets ≥ 100,000 without transfusions and/or exogenous growth factor support (no transfusion or exogenous growth factor within 7 days of assessment);
  2. BM with 5% to 25% blasts and at least a 50% decrease in BM blast percent from baseline;
  3. No evidence of extramedullary disease.
Time Frame: Response was assessed at the completion of the 21-day treatment period of cycles 1, 2, 3.
Population: Intent to Treat Population consisted of all enrolled participants regardless of whether they received lenalidomide.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Participants | 1

5. Secondary Outcome: Number of Participants With a Morphologic CR, CRi, PR or Treatment Failure at Cycles 1, 2 and 3
Description: Disease assessment outcome at the end of Cycles 1-3 based on Cheson criteria:
  Morphologic CR =
  1. ANC ≥ 1000/μL and platelet ≥ 100,000 without transfusions and/or exogenous growth factor support (no transfusion or exogenous growth factor within 7 days of assessment)
  2. BM < 5% blasts evidence of trilineage hematopoiesis
  3. No evidence of extramedullary disease Morphologic CRi =
  1. ANC< 1000/μL and Platelets < 100,000/μL or > 100,000/μL without platelet recovery (requiring transfusion within 7 days of assessment) 2. BM with < 5% blasts and evidence of trilineage hematopoiesis 3. No evidence of extramedullary disease PR =
  1. ANC ≥ 1000/μL and platelets ≥ 100,000 without transfusions and/or exogenous growth factor support
  2. BM with < 5%-25% blasts and at least a 50% decrease in BM blast percent from baseline
  3. No evidence of extramedullary disease Treatment Failure = resistant disease; survival ≥ 7 days post-therapy; failed to achieve CR, CRi, or PR but stable with persistent AML
Time Frame: Response was assessed at the completion of the 21-day treatment period of cycles 1, 2, 3.
Population: The intent to treat population consisted of all enrolled participants regardless of whether they received lenalidomide. Data are reported for participants who began each treatment cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Participants
  Cycle 1 Morphologic CR | 0
  Cycle 1 Morphologic CRi | 0
  Cycle 1 PR | 1
  Cycle 1 Treatment Failure | 13
  Cycle 2 Morphologic CR: number analyzed (Participants) | 8
  Cycle 2 Morphologic CR | 0
  Cycle 2 Morphologic CRi: number analyzed (Participants) | 8
  Cycle 2 Morphologic CRi | 1
  Cycle 2 PR: number analyzed (Participants) | 8
  Cycle 2 PR | 0
  Cycle 2 Treatment Failure: number analyzed (Participants) | 8
  Cycle 2 Treatment Failure | 5
  Cycle 3 Morphologic CR: number analyzed (Participants) | 1
  Cycle 3 Morphologic CR | 0
  Cycle 3 Morphologic CRi: number analyzed (Participants) | 1
  Cycle 3 Morphologic CRi | 1
  Cycle 3 PR: number analyzed (Participants) | 1
  Cycle 3 PR | 0
  Cycle 3 Treatment Failure: number analyzed (Participants) | 1
  Cycle 3 Treatment Failure | 0

6. Secondary Outcome: Number of Participants Who Received a Haematopoietic Stem Cell Transplant (HSCT)
Description: The number of participants who had undergone a haematopoietic stem cell transplant was calculated over the total number of participants in the ITT population. Percentages were also calculated based on whether the transplantation was the first, second, or subsequent transplant post IP administration.
Time Frame: From first dose of study drug up to 5 years post HSCT
Population: The intent to treat population consisted of all enrolled participants regardless of whether they received lenalidomide.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Participants
  Any Transplant After Treatment Start | 2
  First Transplant After Treatment Start | 2
  Second Transplant After Treatment Start | 0
  Any Subsequent Transplant After Treatment Start | 0

7. Secondary Outcome: Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAE)
Description: A TEAE was defined as any adverse event (AE) occurring or worsening on or after the first treatment of lenalidomide and within 28 days after the last dose. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.3 and based on the following scale: Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death.
Time Frame: From the first dose of study drug until 28 days after the last dose of study drug; up to data cut off date of 31 December 2017; maximum duration of treatment was 12 weeks
Population: The safety population consisted of all participants who received at least one dose of lenalidomide.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Participants
  Any TEAE | 17
  Any TEAE Related to Lenalidomide | 15
  Any Grade 3/4 TEAE | 17
  Any Grade 3/4 TEAE Related to Lenalidomide | 11
  Any Grade 5 TEAE | 1
  Any Serious TEAE | 13
  Any Serious TEAE Related to Lenalidomide | 5
  Any Serious TEAE Leading to Dose Discontinuation | 3
  Any TEAE Leading to Dose Discontinuation | 3
  Any TEAE Leading to Dose Reduction | 4
  Any TEAE Leading to Dose Interruption | 7
  Any TEAE Leading to Death | 1

8. Secondary Outcome: Percentage of Participants With of Graft Versus Host Disease (GVHD)
Description: Acute graft versus host disease generally occurs after allogeneic hematopoietic stem cell transplantation. It is a reaction of donor immune cells against host tissues. The 3 main tissues that acute GVHD affects are the skin, liver, and gastrointestinal tract. Chronic GVHD is scored per the National Institute of Health consensus conference grading system. Clinical manifestations of chronic GVHD include skin involvement resembling lichen planus or the cutaneous manifestations of scleroderma; dry oral mucosa with ulcerations and sclerosis of the gastrointestinal tract; and a rising serum bilirubin concentration.
Time Frame: From the first dose of study drug to 28 days after the last dose of study drug; up to data cut off date of 31 December 2017; maximum treatment was 12 weeks
Population: The Safety population consisted of all participants who received at least 1 dose of lenalidomide.
Measure: Number; unit: Percentage of Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Percentage of Participants | 0

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration of Lenalidomide (AUC-t)
Description: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration, calculated by linear trapezoidal method when concentrations were increasing and the logarithmic trapezoidal method when concentrations were decreasing.
Time Frame: Pharmacokinetic (PK) sampling was conducted after lenalidomide administration at Cycle 1 and was weight dependent at these timepoints: 0.5, 1, 2, 4, 6, 8 and 24 hours. The 24 hour PK sample was taken prior to the lenalidomide dose on Day 2.
Population: The pharmacokinetic population included participants who received at least one dose of lenalidomide and had at least one measurable lenalidomide concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
ng*h/mL | 5378.83 (57.3)

10. Secondary Outcome: Area Under the Plasma Concentration Time Curve From 0 Extrapolated to Infinity (AUC-inf, AUC0∞) Of Lenalidomide
Description: Area under the plasma concentration-time curve from time 0 extrapolated to infinity, calculated as [AUCt + Ct/ λz]. Ct is the last quantifiable concentration. No AUC extrapolation was performed with unreliable λz.
Time Frame: Pharmacokinetic sampling was conducted after lenalidomide administration at Cycle 1 and was weight dependent at these timepoints: 0.5, 1, 2, 4, 6, 8 and 24 hours. The 24 hour PK sample was taken prior to the lenalidomide dose on Day 2.
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
ng*h/mL | 5656.67 (52.8)

11. Secondary Outcome: Maximum Observed Concentration (Cmax) of Lenalidomide
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: PK sampling was conducted after lenalidomide administration at Cycle 1 and was weight dependent at these timepoints: 0.5, 1, 2, 4, 6, 8 and 24 hours. The 24 hour PK sample was taken prior to the lenalidomide dose on Day 2.
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
ng/mL | 1252.08 (43.8)

12. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Lenalidomide
Description: Time to cmax was obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 11
Population: as for outcome 9
Measure: Median (Full Range); unit: Hours
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Hours | 2.000 [0.5500 to 4.000]

13. Secondary Outcome: Terminal Half-Life (t1/2) of Lenalidomide
Description: Terminal phase half-life in plasma, calculated as [(ln 2)/λz]. Terminal half-life was only calculated when a reliable estimate for λz could be obtained.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
hours | 2.311 (43.3)

14. Secondary Outcome: Apparent Total Clearance (CL/F) of Lenalidomide
Description: Apparent volume of distribution, calculated as [(CL/F)/λz].
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml/min
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
ml/min | 172.09 (52.5)

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Lenalidomide
Description: Apparent volume of distribution, calculated as [(CL/F)/λz].
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
Liters | 34.42 (57.0)

16. Secondary Outcome: Correlation of Peripheral White Blood Cell Count, Absolute Blast Count and Cytogenetics With Response to Lenalidomide
Description: Correlation of peripheral white blood cell count, absolute blast count and cytogenetics with response to lenalidomide was not performed since only 1 participant met the primary efficacy endpoint of morphological CR/CRi, and due to scarcity of relevant data, it was not practical or meaningful to analyze to perform the analysis on blood counts and response to lenalidomide.
Time Frame: Not Performed
Population: Due to scarcity of relevant data, it was not practical or meaningful to analyze or perform the analysis on blood counts and response to lenalidomide.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the date of the first dose of lenalidomide until 28 days after the last dose of lenalidomide; up to the date the last patient discontinued follow-up 11 January 2019; maximum treatment duration was 12 weeks.
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 13/17
Serious Adverse Events (participants affected / at risk) | 13/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Cellulitis (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=17)
Anaemia (Blood and lymphatic system disorders) | 10
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Splenic infarction (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 4
Hypoacusis (Ear and labyrinth disorders) | 1
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Neutropenic colitis (Gastrointestinal disorders) | 1
Oral mucosal erythema (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Catheter site haematoma (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 7
Hepatosplenomegaly (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Sinusitis (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 4
Anti-platelet antibody positive (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 4
Blood fibrinogen decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 1
International normalised ratio increased (Investigations) | 3
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Fluid overload (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Lethargy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Device issue (Product Issues) | 1
Device occlusion (Product Issues) | 1
Thrombosis in device (Product Issues) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Phonophobia (Psychiatric disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The results of the efficacy analysis were reviewed by an independent Data Monitoring Committee, which concluded that the study would not proceed to Stage 2, given that the efficacy criteria for continuation of the study to Stage 2 had not been met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 30 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 60 additional days. Investigator must delete confidential data before submission or defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT02538965/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT02538965/SAP_001.pdf